CLINICAL TRIAL: NCT00925496
Title: Patient Benefit From the New Modular Shoulder Prosthesis PROMOS - a Multicentre Cohort Study
Brief Title: Patient Benefit From the New Modular Shoulder Prosthesis PROMOS
Acronym: Promos
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: D10054
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Primary or Secondary Omarthrosis of the Shoulder Joint
Keywords: Omarthrosis shoulder joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard PROMOS prosthesis: Patients receiving a standard PROMOS prosthesis
- Reverse PROMOS prosthesis: Patients receiving a reverse PROMOS prosthesis

SUMMARY:
Overall study design:

This study is a prospective, non-randomized, multicenter postmarket clinical follow-up study with two study arms using the two shoulder prosthesis PROMOS™ STANDARD (group A) and PROMOS REVERSE™ (group B). The study will collect efficacy and safety data over 10 years.

DETAILED DESCRIPTION:
Primary objective of the study:

The primary objective is to quantify patient benefit after primary total shoulder arthroplasty with the modular PROMOS™ shoulder system in a multicenter cohort study (real world approach). Patient benefit will be quantified using objective and validated subjective measures of function, activities of daily living (ADL) and quality of life (QoL).

Secondary objectives:

* Rate of implant related findings like radiological loosening of the glenoid and complications like intraoperative stem fissures
* Prosthesis survival at common time points, e.g. 5 and 10 years

ELIGIBILITY:
Eligibility:

* Ages eligible for study: minimal age of 18 years
* Genders eligible for study: both
* Accepts healthy volunteers: no

Inclusion Criteria:

* Primary or secondary omarthrosis as an indication for primary total shoulder arthroplasty
* Massive rotator cuff rupture
* Willing an able to give written informed consent to participate in the study including follow-ups

Exclusion Criteria:

* Previous ipsilateral shoulder arthroplasty (group A and B)
* Late stage rotator cuff disease (only group A)
* Acute shoulder trauma (group A and B)
* General medical contraindication to surgery (group A and B)
* Legal incompetence (group A and B)
* Tumour / malignoma (group A and B)
* Recent history of substance abuse (group A and B)
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder) (group A and B)
* Known hypersensitivity to the materials used (group A and B)
* Bacterial infection at the time point of operation (group A and B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2009-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures: Patient benefit will be measured with the SPADI and Constant Murley score at the joint level, with the QuickDASH for the upper extremity and the SF-36 mental score as a generic tool. | Preop / 6M / 1Y / 2Y / 5Y / 10Y

SECONDARY OUTCOMES:
Active and passive ROM and strength / Rate of implant related complications / Rate of implant related findings like radiological loosening of the glenoid / Prosthesis survival at common time points, e.g. 5 and 10 years | Preop / 6M / 1Y / 2Y / 5Y / 10Y

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Kaspar Schwyzer, Dr. med., Principal Investigator — Schulthess Klinik
Locations (2):
- Orthopaedische Praxis / Praxisklinik, Münster, Germany
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided